CLINICAL TRIAL: NCT06629480
Title: Incidence of Metabolic Syndrome in People Living With HIV Without ExperienCe to ART Who Start DoLutegravir Based-Regimen Compared With BictegrAvir Based-RegimeN After 48 Weeks (MICTLAN Trial)
Brief Title: Incidence of Metabolic Syndrome in People Living With HIV Without ExperienCe to ART Who Start DoLutegravir Based-Regimen Compared With BictegrAvir Based-RegimeN
Acronym: MICTLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, José Antonio Mata Marín, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2021-3502-084
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Antiretroviral Treatment; HIV Infection; Metabolic Cardiovascular Syndrome
Keywords: Weight gain; Metabolic syndrome; Dyslipidemia
MeSH Terms: conditions — HIV Infections; Metabolic Syndrome; Weight Gain; Dyslipidemias | interventions — bictegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIC/TAF/FTC (Active Comparator)
  Interventions: Drug: Bictegravir
- DTG/ABC/3TC (Active Comparator)
  Interventions: Drug: Bictegravir

INTERVENTIONS:
Drug: Bictegravir — The aim of the study was to identify the incidence of MetS at 48 weeks for ATP III score in patients living with HIV (PLH) who started antiretroviral therapy (ART) with Dolutegravir based-regimen compared with Bictegravir based-regimen. A randomized open clinical trial was developed with men PLH who started ART randomized to BIC/FTC/TAF or DTG/3TC/ABC.

SUMMARY:
The aim of the study was to identify the incidence of MetS at 48 weeks for ATP III score in patients living with HIV (PLH) who started antiretroviral therapy (ART) with Dolutegravir based-regimen compared with Bictegravir based-regimen. MICTLAN is a randomized open clinical trial developed with men PLH who started ART randomized to BIC/FTC/TAF or DTG/3TC/ABC. Weight, height, blood pressure, and waist circumference and electriccircumference were measured during routine clinical care; in addition, electric bioimpedance were measured atmeasuredwas done; repeated measures of weight in kilograms were done at baseline, 24 and 48 weeks. Metabolic laboratory tests were done on each visit.

DETAILED DESCRIPTION:
The aim of this study was to compare the incidence of MetS at 24 weeks by ATP III score in PLHpatients living with HIV who started antiretroviral therapy (ART) with Dolutegravir based-regimen vs. Bictegravir based-regimen. An open-label randomized clinical trial was conducted,from February 2021 through December 2022, in HIV clinic at the national medical center "La Raza", Mexico city. the primary endpoint was the incidence of MetS at 48 weeks comparing BIC/FTC/TAF with DTG/3TC/ABC in patients with HIV type 1 (HIV-1) infection starting ART.Study subjects were men who have sex with men (MSM) with HIV-1 infection ≥18 years old, living with HIV, naïve to ART (PLHIV). The trial enrolled residents of Mexico City and Mexico State from February 2021 through February 2024. Inclusion criteria were men over ≥18 years , a viral load of at least of 500 copies/ or more per milliliter, and a creatinine clearance over 60 ml/ per minute (CKD-EPI formula). Among the exclusion criteria were MetS, comorbidities or prescription of drugs associated with weight gain or weight loss or current treatment for tuberculosis. Each patient received a personalized eating plan based on the equivalent food system method adjusted to their energy requirements before starting treatment by a nutritionist . The primary endpoint was the incidence of MetS at week 24. Secondary objectives were the percentage of patients with an HIV-1 RNA level of less than 40 copies/ per mlilliliter, CD4+ count changes, and side-effect profile and safety, including findings on physical examination and laboratory analyses. Body composition was measured at baseline and at 24 weeks using a next generation bioimpedance device. Each patient was measured in duplicate to ensure better results and to avoid minimal changes. An ultrasonography (US) to measure visceral and subcutaneous fat was donemeasured. Waist circumference was also measured in the fasting state by using a non-retractable material flexible ruler. There was no testing of HIV resistance at screening. Patients with two confirmed elevations in the HIV-1 RNA level to 1000 copies or more per milliliter after week 24 were tested for drug resistance, together with their stored baseline samples. Weight and height were measured every medical visitduring routine clinical care, and recorded in electronic health records. Repeated measures of weight in kilograms (kg) were done at baseline 24 and 48 weeks. Descriptive results were summarized using median and interquartile range (IQR). Percentage was obtained in order to evaluate the weight gain classification. The main outcome variable was the incidence of MS at 48 weeks. We assessed weight change and metabolic changes at 48 weeks with a Wilcoxon signed-rank test. Mann Whitney U-test was used to compare between groups of INSTI. The effectiveness outcomes were analyzed in the intention-to-treat population and the safety outcomes were analyzed in the as-treated population. All analyses were conducted using SPSS software (version 29; SPSS IBM Corp., Armonk, NJ, USA)

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men (MSM) with HIV-1 infection
* ≥18 years old
* Living with HIV
* Naïve to ART
* Creatinine clearance over 60 ml/ per minute (CKD-EPI formula)

Exclusion Criteria:

* Metabolic Syndrome
* Comorbidities or prescription of drugs associated with weight gain or weight loss
* Current treatment for tuberculosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Metabolic Syndrome | 48 weeks
  Incidence of MetS at 48 weeks for ATP III score in patients living with HIV (PLH) who started antiretroviral therapy (ART) with Dolutegravir based-regimen compared with Bictegravir based-regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Infectología, "La Raza" National Medical Center, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided